CLINICAL TRIAL: NCT04147949
Title: Randomized, Double-Blind, Placebo-Controlled, Crossover, Proof-of-Concept Phase 2 Study to Test Efficacy and Safety of AV-101 (L-4-chlorokynurenine) in Parkinson's Disease Subjects With Levodopa-Induced Dyskinesia
Brief Title: AV-101 (L-4-chlorokynurenine) in Parkinson's Disease Subjects With Levodopa-Induced Dyskinesia
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: VistaGen Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: VSG-CL-004
Record Dates: First submitted 2019-10-27; First posted 2019-11-01 (Actual); Last update posted 2021-05-26 (Actual); Status verified 2021-05

CONDITIONS: Parkinson Disease; Dyskinesia, Medication-Induced; L-Dopa Causing Adverse Effects in Therapeutic Use
MeSH Terms: conditions — Parkinson Disease; Dyskinesia, Drug-Induced

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- AV-101 (Experimental): 1440 mg of L-4-chlorokynurenine administered twice a day orally
  Interventions: Drug: AV-101
- Placebo (Placebo Comparator): Matching capsules of placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AV-101 — Oral capsules taken twice daily for 14 days
  Other Names: L-4-chlorokynurenine
  Arms: AV-101
Drug: Placebo — Oral capsules taken twice a day for 14 days
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled, crossover, proof-of-concept Phase 2 study to test efficacy and safety of AV-101 (L-4-chlorokynurenine) in Parkinson's Disease subjects with levodopa-induced dyskinesia. The trial will be conducted in two treatment periods, in which each treatment period will consist of 14 days. The two treatment periods will be separated by a 1-week washout period. During the first treatment period, subjects meeting all eligibility criteria will be randomly assigned to receive either 1440 mg AV-101 or placebo in a 1:1 ratio. AV-101 or placebo will be administered BID for 14 days (every 12 hours). After the washout period, all subjects will be crossed over to receive the alternate treatment during the second treatment period (14-day period).

On the last day of each treatment period (Visit 4 [Day 14] and Visit 7 [Day35]), subjects will be assessed in clinic while in the practically "off" state and will receive the morning dose of the study drug at the clinic. This will be followed, within 25-30 minutes, by oral administration of a dose of levodopa that is 150% of the subject's normal dose. Assessments of dyskinesia and PD motor symptoms will be performed before and after levodopa/carbidopa administration.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female adults, 30 to 80 years of age, inclusive.
2. Diagnosis of idiopathic PD meeting the United Kingdom Parkinson's disease Society Brain Bank criteria.
3. Levodopa-induced dyskinesia present greater than 25% of the day as per MDS-UPDRS.
4. Dyskinesia of at least moderate severity as per MDS-UPDRS
5. Subjects currently receiving anti-parkinsonian medications that contain levodopa and carbidopa are eligible provided they have been on a stable dose of these medications for at least 1 month prior to randomization.
6. Subjects currently receiving antidepressants such as selective serotonin reuptake inhibitors, provided the dose has been stable for at least 1 month prior to randomization.
7. If female, a status of non-childbearing potential or use of an acceptable form of birth control per the following specific criteria:

   1. Non-childbearing potential (e.g., physiologically incapable of becoming pregnant, i.e., permanently sterilized (status post hysterectomy, bilateral tubal ligation), or is postmenopausal with her last menses at least 1 year prior to screening); or
   2. . Childbearing potential, and meets all of the following criteria: i. Women with a negative urinary pregnancy test at screening, confirmed by a negative urinary pregnancy test at randomization prior to receiving study treatment.

ii. Women who are willing and able to continuously use one of the following methods of birth control during the course of the study, defined as those which result in a low failure rate (i.e., less than 1% per year) when used consistently and correctly: implants, injectable or patch hormonal contraception, oral contraceptives, intrauterine device, sexual abstinence. The form of birth control will be documented at screening.

iii. Male partner must use a condom.

Exclusion Criteria:

1. Women with childbearing potential who are not willing to use one of the specified forms of birth control during the study or whose partner is unwilling to use a condom.
2. Women who are pregnant or breastfeeding.
3. Women with a positive pregnancy test at screening or baseline.
4. Currently taking a prohibited adjunct therapy such amantadine or monoamine oxidase (MAO) inhibitors must be discontinued at least 3 weeks prior to baseline.
5. Subject had a prior surgery for PD except Deep Brain Stimulation (Deep Brain Stimulation must not have been performed within one year of screening)
6. Hoehn and Yahr score of 5 when "off".
7. Subject with Cognitive impairment and/or history of psychiatric manifestations or active hallucinations.
8. History of positive screening urine test for drugs of abuse at screening: cannabinoids (if the subject has a legitimate medical prescription for cannabis, subject must agree to abstain during the entirety of the study and to have a negative test at baseline), cocaine, barbiturates, opiates. A positive benzodiazepine result will be allowed if there is a valid and prescribed medical use for these agents. For all other positive results, a single re-test is permitted at the judgement of the investigator; results of any retest must be available prior to the baseline visit and must be negative.
9. In poor general health, as ascertained by medical history, physical examination (including measurement of vital signs), clinical laboratory evaluations, and 12-lead electrocardiogram (ECG).

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-08 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Unified Dyskinesia Rating Scale | 14 days
  (UDysRS) Part 3 AUC
Unified Dyskinesia Rating Scale | 14 days
  (UDysRS) Part 3 Peak Score

SECONDARY OUTCOMES:
Movement Disorder Society- Unified Parkinson's Disease Rating Scale | 14 days
  (MDS-UPDRS) part III (Parkinsonian disability)

IPD SHARING:
Plan to Share IPD: No